CLINICAL TRIAL: NCT05691686
Title: Effects of Less-processed Whole Grain Bread Products (Wheat and Fortified With Legumes) on Postprandial Glucose and Subsequent Metabolic Responses.
Brief Title: Bread Structure and Postprandial Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Amalia Yanni, Research and Teaching Associate, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 513.26-07-2021
Record Dates: First submitted 2022-12-22; First posted 2023-01-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-01

CONDITIONS: Postprandial Hyperglycemia
Keywords: bread; food structure; glycemic control; appetite regulation
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Finely milled whole wheat-legume bread (Experimental): Treatment with finely milled whole wheat-legume bread.
  Interventions: Other: Finely milled whole wheat-legume bread
- Less processed whole wheat-legume bread (Experimental): Treatment with less processed whole wheat-legume bread.
  Interventions: Other: Less processed whole wheat-legume bread
- Less processed whole wheat bread (Experimental): Treatment with of less processed whole wheat bread.
  Interventions: Other: Less processed whole wheat bread
- Reference Food (white wheat bread) (Active Comparator): Treatment with reference food.
  Interventions: Other: White wheat bread

INTERVENTIONS:
Other: Finely milled whole wheat-legume bread — The intervention examines the effect of finely milled wheat-legume bread in subjects with normal body weight.
  Arms: Finely milled whole wheat-legume bread
Other: Less processed whole wheat-legume bread — The intervention examines the effect of less processed whole wheat-legume bread in subjects with normal body weight.
  Arms: Less processed whole wheat-legume bread
Other: Less processed whole wheat bread — The intervention examines the effect of less processed whole wheat bread in subjects with normal body weight.
  Arms: Less processed whole wheat bread
Other: White wheat bread — The intervention examines the reference food product in subjects with normal body weight.
  Arms: Reference Food (white wheat bread)

SUMMARY:
The structural properties of bread are considered one of the most important factors that can affect its digestibility, glucose homeostasis and postprandial metabolic responses. The purpose of this study is to examine the effects of consumption of less processed whole grain bread products (wheat and fortified with legumes) in comparison with finely milled whole grain bread products on postprandial glycaemic response and appetite regulation.

DETAILED DESCRIPTION:
Postprandial glucose response caused by bread products of different degree of processing, as well as their appetite regulating properties will be evaluated. In the intervention there are totally four samples, the reference (white wheat bread), the less processed whole wheat bread, the whole wheat bread fortified with finely milled legumes (chickpeas), the whole wheat bread fortified with less processed legumes (chickpeas). The volunteers that will be enrolled in the study should be apparently healthy subjects (women and men) with normal body weight. Certain effects related to the structure of the different products on glycemic and insulinemic responses, subjective appetite ratings and other parameters will be examined.

ELIGIBILITY:
Inclusion Criteria:

* normal exercise and dietary habbits
* weight stable for at least 3 months before enrollment

Exclusion Criteria:

* pregnancy and lactation
* diabetes
* chronic medical illness
* regular intense exercise (>5 hrs/week)
* alcohol consumption >2 drinks/day

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in glucose incremental area under the curve (iAUC) after consumption of the breads compared to the iAUC after consumption of the reference food. | Time points: 0 (before food consumption), 30, 45, 60, 90,120,180 minutes postprandially (4 times in total).
  Blood glucose concentration will be measured for each participant before and after the test foods, with blood samples being collected at specific time points: 0 (before food consumption), 30, 45, 60, 90, 120, 180 minutes postprandially for each food.

SECONDARY OUTCOMES:
Subjective appetite ratings | Time points: 0 (before food consumption), 30, 60, 90,120,180 minutes postprandially (4 times in total).
  Subjective evaluation of hunger, satiety, and desire to eat with Visual Analogue Scales, before the consumption and 30, 60, 90, 120, 180 minutes after (0-100 mm with 0 indicating no hunger or perceived ability to consume food/no satiety or no fullness). Difference in perception of these parameters will be measured and compared between the experimental condition and the control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Tentolouris, Professor, Study Chair — National and Kapodistrian University of Athens; Vaios Karathanos, Professor, Study Chair — Harokopio University of Athens
Locations (1):
- Amalia Yanni, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No